CLINICAL TRIAL: NCT00164541
Title: An Arts-Based Initiative for the Prevention of Violence Against Women and Girls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3292; US4/CCU319009
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Violence
Keywords: dating violence; violence against women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Arts Based Program
Behavioral: Curriculum

SUMMARY:
this project will evaluate a community and school based program to promote healthy relationships and prevent violence (physical, emotional and sexual dating violence) among predominately African American middle school adolescents in an urban setting (Baltimore, MD).

DETAILED DESCRIPTION:
This initiative includes 4 major components: 1) A variety of arts based student activities related to violence prevention (during and after school theatre projects, during and/or after school visual arts project, and the web page design project. (All students will either directly participate in these activities or at least see them), 2) Curricular components for all 7th graders, 3) Violence prevention and early intervention student support/discussion groups, and 4) Faculty and staff training on the subject. The evaluation is a quasi-experimental pre/post test comparison group design (2 schools in each group), where our comparison schools convert to intervention schools one year after serving as comparison schools. We are using both group (student and teacher surveys) and school wide (climate of the school) measures pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students in four middle schools in urban Baltimore, MD (Dunbar, Lombard, Calverton and Lemmel Middle Schools)

Exclusion Criteria:

-

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1440 (Actual)
Dates: Start 2004-09; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Dating violence perpetration | past 12 months

SECONDARY OUTCOMES:
Dating violence victimization | past 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline Campbell, PhD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Dunbar Middle School, Baltimore, Maryland
  - Calverton, Baltimore, Maryland
  - Lemmel Middle School, Baltimore, Maryland
  - Lombard School, Baltimore, Maryland